CLINICAL TRIAL: NCT02597621
Title: Biomarkers for Therapy Response in Drug-resistant Tuberculosis
Status: Completed | Type: Observational
Sponsor: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Christoph Lange, Head of International Health / Infectious Diseases, University Lübeck, Research Center Borstel
Other Study IDs: M/XDR_BIO_01
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Multidrug-resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- M/XDR: The M/XDR-cohort will consist of patients with a suspected infection with an M/XDR-TB strain.The suspicion will be held on behalf of molecular biological methods (i.e. GeneXpert, detection of rifampicin resistance with high probability of simultaneous isoniazid resistance). The suspected cases will be confirmed by culture (n= 20). Empirically, less than 10% of the cases have an XDR-TB
  Interventions: Other: no intervention
- Susceptible: The non M/XDR-TB cohort will consist of patients with no suspected infection with an M/XDRTB strain. The suspicion will be out ruled on behalf of molecular biological methods (i.e.GeneXpert, detection of rifampicin resistance with high probability of simultaneous isoniazid resistance). The non M/XDR-TB cases will be confirmed by culture (n= 20). Empirically, about 90% of these patients have no drug resistance against first line drugs.
  Interventions: Other: no intervention
- Healthy Controls: Healthy controls.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Multi-center, observational, prospective cohort study including patients with multidrug-resistant tuberculosis at different sites in Germany.

The aim the study is the identification of biomarkers for therapy response.

DETAILED DESCRIPTION:
The increasing rates of multidrug-resistant (MDR) tuberculosis (TB) are causing great concern. The current study that will be conducted at different centers in Germany. Biomarkers for treatment response during the course of the tuberculosis therapy will be evaluated. The study will be conducted with funding of the German Center for Infection Research (DZIF).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed pulmonary MDR-TB
* Subject able and willing to give informed consent

Exclusion Criteria:

* HIV infection
* physical or mental inability preventing study participation at the discretion of the investigator
* member of a vulnerable or special population (prisoner, soldier, mentally ill, under guardianship)
* age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with microbiologically confirmed pulmonary MDR-TB
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Identification of biomarkers for therapy response | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Borstel, Borstel, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Heyckendorf J, Marwitz S, Reimann M, Avsar K, DiNardo AR, Gunther G, Hoelscher M, Ibraim E, Kalsdorf B, Kaufmann SHE, Kontsevaya I, van Leth F, Mandalakas AM, Maurer FP, Muller M, Nitschkowski D, Olaru ID, Popa C, Rachow A, Rolling T, Rybniker J, Salzer HJF, Sanchez-Carballo P, Schuhmann M, Schaub D, Spinu V, Suarez I, Terhalle E, Unnewehr M, Weiner J 3rd, Goldmann T, Lange C. Prediction of anti-tuberculosis treatment duration based on a 22-gene transcriptomic model. Eur Respir J. 2021 Sep 2;58(3):2003492. doi: 10.1183/13993003.03492-2020. Print 2021 Sep. PMID 33574078